CLINICAL TRIAL: NCT06194357
Title: Developing an Integrated Mindfulness-based Health Qigong Intervention (iMBHQ) for COVID-19 Survivors and Caregivers to Improve Their Physical and Psychological Wellness
Brief Title: Integrated Mindfulness-based Health Qigong Intervention for COVID-19 Survivors and Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Chair Professor and Head of Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KW/EX-23-001(179-01)
Record Dates: First submitted 2024-01-04; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Infection
Keywords: COVID-19 Survivors; caregivers; mindfulness-based health Qigong intervention; physical wellness; psychological wellness
MeSH Terms: conditions — COVID-19; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will receive training on Qigong exercise and mindfulness.
  Interventions: Other: Mindfulness-based Health Qigong Intervention
- Control group (No Intervention): Control group will not receive intervention.

INTERVENTIONS:
Other: Mindfulness-based Health Qigong Intervention — Participants are introduced the practice of the most essential skills, particularly mindfulness, the basic movements of Qigong and the use of the resources package. Following the initial session, participants will kick off 8 bi-weekly online sessions of Mindfulness-based interventions approximately two hours each via the Mobile App. Afterwards, participants will be asked to practice Qigong for 30 minutes per day with five days weekly for another 8 weeks. Follow-up sessions will be conducted by an experienced coach via the Mobile App. After the first 16-week intervention, booster sessions will be provided every 3 months to revise the interventions and follow-up assessments will be completed every 6 months for 2 years.
  Arms: Intervention group

SUMMARY:
COVID-19-related depression, anxiety, and stigma are expected to have short-term and long-term adverse impacts on mental health, help seeking and preventive behaviours in affected individuals, including care providers and the general population. Health qigong (HQ), a form of traditional Chinese martial arts with emphasis placed on the body movement and status of mind, has been demonstrated to enhance both physical and mental health. Mindfulness-based interventions (MBIs), another mind-body treatment, have become increasingly popular for treating a number of health problems. This study proposes an integrated intervention that combines the effects of HQ and MBIs (iMBHQ) to improve the mental wellbeing of COVID-19 survivors, caregivers including healthcare providers and family members as well as the general public in the community.

DETAILED DESCRIPTION:
Objective:

The study aims to examine whether iMBHQ can improve the physical and psychological wellness of COVID-19 survivors, caregivers and the general public in the community.

Procedures:

Participants will be randomized into either the treatment group (16-week iMBHQ program) or the control group. For the treatment group, a face-to-face initial session will be arranged for each participant to introduce the practice of the most essential skills, particularly mindfulness, the basic movements of Qigong and the use of the resources package. Following the initial session, participants will kick off 8 bi-weekly online sessions of MBIs approximately two hours each via the Mobile App. Afterwards, participants will be asked to practice Qigong for 30 minutes per day with five days weekly for another 8 weeks. Follow-up sessions will be conducted by an experienced coach via the Mobile App. After the first 16-week intervention, booster sessions will be provided every 3 months to revise the interventions and follow-up assessments will be completed every 6 months for 2 years.

Participants:

will be asked to practice Qigong for 30 minutes per day with five days weekly for another 8 weeks. Follow-up sessions will be conducted by an experienced coach via the Mobile App. After the first 16-week intervention, booster sessions will be provided every 3 months to revise the interventions and follow-up assessments will be completed every 6 months for 2 years.

Results:

The investigators predict that the integrated intervention developed will significantly reduce fear, anxiety and stigma in COVID-19 survivors, their caregivers and the general public by improving stress, cognitive, and mood coping strategies.

Conclusions:

The findings will be able to explain the effects and outcomes of integrated intervention derived from the hypothetical model which the investigators will propose. The outcomes will also help transform the hypothetical model into a psychosocial and rehabilitation theory, which can explain many of the psychosocial and behavioral consequences that may hinder the recovery of those affected by COVID-19 and hinder their caregivers and the general public to seek help and take preventive measures against the disease. The findings will also demonstrate that the integrated intervention developed by the research group will be the long-term and cost-effective rehabilitation management approaches for COVID-19 survivors, caregivers, and the general public to promote their physical and psychological wellbeing in the community

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 survivors: people aged 18 years or above who were infected by COVID-19 (both symptomatic and asymptomatic) and clinically recovered
* Caregivers of COVID-19 patients, including family members or medical professionals who have contacts with patients diagnosed COVID-19 aged 18 years or above
* General healthy public aged 18 years or above

Exclusion Criteria:

* people diagnosed severe and/or chronic conditions that prevent the practice of Qigong (e.g., acute exacerbation of dyspnoea, severe cardiopulmonary disease) or mindfulness intervention,
* people with severe psychiatric disorder
* people who have regular psychiatric follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Psychological wellbeing | 2 years
  Depression, Anxiety and Stress Scale (DASS-12)

SECONDARY OUTCOMES:
Multidimensional Assessment of Interoceptive Awareness (MAIA) | 2 years
  12-item Short Form healthy survey (SF-12); Rumination Reflection Questionnaire (RRQ); Hyperarousal Scale COVID-19 Fear Scale; Stigma: Perceived stigma and Self-stigma Scale; Attitudes toward rapid testing and vaccine scale

CONTACTS AND LOCATIONS:
Overall Officials: Wing Hong, Hector TSANG, Prof, Principal Investigator — Department of Rehabilitation Science, Faculty of Health and Social Sciences
Locations (1):
- Princess Margaret Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No